CLINICAL TRIAL: NCT03968731
Title: Meibomian Gland Dysfunction Management With Zocular Eyelid System Treatment (ZEST) to Relieve Contact Lens Discomfort
Brief Title: Meibomian Gland Dysfunction Management With ZEST Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Incarnate Word (Other)
Responsible Party: Principal Investigator, SRIHARI NARAYANAN, Professor, University of the Incarnate Word
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-05-007
Record Dates: First submitted 2019-05-28; First posted 2019-05-30 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Meibomian Gland Dysfunction; Dry Eye Syndromes; Ocular Surface Disease
Keywords: contact lens discomfort
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ZEST treatment (Experimental): The study subjects will receive the ZEST treatment protocol (Zocular Eyelid System treatment) to treat Meibomian Gland Dysfunction causing Contact Lens discomfort symptoms.
  Interventions: Other: Zocular Eyelid System Treatment

INTERVENTIONS:
Other: Zocular Eyelid System Treatment — Zocular products contain okra-infused Zocusome micelles that gently lift and clear the oil, debris, and residue on eyelid margins. THerefore, the ZEST treatment is expected to improve signs and symptoms of Meibomian gland dysfunction (MGD) and reduce Contact lens discomfort associated with MGD.
  Other Names: ZEST

SUMMARY:
The purpose of this study is to investigate if cleaning the eyelid margin with the ZEST protocol (Zocular Eyelid System Treatment) in patients intolerant to contact lens wear consequent to Meibomian gland dysfunction (MGD) will improve the MGD and contact lens wear comfort.

DETAILED DESCRIPTION:
Meibomian gland dysfunction (MGD) is a common clinical condition seen in optometric practices that affects the quality of the tear fluid on the surface of the eye. In MGD, the Meibomian glands secrete lipids which are of poor quality and altered composition. This results in a dysfunctional tear fluid causing symptoms of ocular irritation (such as dry eyes). Patients who use contact lenses on a daily basis suffer from contact lens intolerance due to their MGD.

A study done by Korb and Blackie in 2013 demonstrated that manual debridement of the lid margin using a spatula is a viable management option for MGD and blepharitis. The investigators of this proposed study have researched the effect of debridement of lid debris (Either electronic debridement with BlephEx or manual debridement using a golf spud) in relieving signs and symptoms of blepharitis (which comprises MGD as well) in patients who do not wear contact lenses on a daily basis as well as in patients who wear contact lenses on a daily basis. The investigators obtained positive results from those studies. Signs and symptoms of MGD and Blepharitis improved in patients following lid margin debridement treatments. The ZEST protocol offers an alternate paradigm for cleaning the eyelid margins. The Zocular products contains okra-infused Zocusome micelles that gently lift and clear the oil, debris, and residue on eyelid margins Presumably, the ZEST treatment protocol will benefit patients who use contact lenses on a daily basis and suffer from symptoms of lens intolerance, since similar treatment / cleaning of lid margin debris has shown to be beneficial for these patients.

Therefore, this study will investigate if the ZEST protocol can relieve symptoms of contact lens intolerance caused by MGD.

There are no clinical studies using the ZEST protocol for the betterment of contact lens comfort in patients who have MGD. Hence, the proposed study will provide new and useful information about this treatment option for managing contact lens intolerance due to MGD. The data generated will directly benefit clinical practice and impact several millions of patients who suffer from intolerance to contact lens wear due to MGD.

ELIGIBILITY:
Inclusion Criteria:

* Clinically determined presence of Meibomian gland dysfunction
* Patient Self-reported discomfort with contact lens wear
* Use of contact lenses on a daily basis

Exclusion Criteria:

* Subjects should not be under active medical treatment for MGD or Blepharitis (inflammation of the eyelid margins) as this will negate the effects of the treatment offered in the proposed study.
* Subjects should not be using prescription eye drops for any reason. Subjects should not be taking any systemic Anti-inflammatory or anti-biotic medication during the course of the study as these medications can alter the effects of the treatment offered in the proposed study.
* Subjects should not have received any form of eyelid margin debridement (such as BlephEx or Manual debridement or ZEST treatment) in the sixty days prior to start of the study as the study treatment will be redundant and no benefits may be perceived by the subject.
* Subjects cannot participate in this study if they are allergic to Okra or Okra-based products (since Zocular products contain an extract from the Okra plant).

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Contact Lens Questionnaire score | One month
  Contact Lens Dry Eye Questionnaire score (CLDEQ-8) ranging from 0 to 41 points. A score of zero points on the CLDEQ-8 will mean the patient is completely asymptomatic whereas a score of 41 points will mean the patient is highly symptomatic for Contact Lens discomfort.
Dry Eye Questionnaire score | One month
  Ocular Surface Disease Index (OSDI) score ranging from 0 to 48 points. A score of zero on the OSDI will mean the patient does not have any dry eye symptoms whereas a score of 48 will mean that the patient is highly symptomatic for dry eye.

SECONDARY OUTCOMES:
MMP-9 expression | One month
  Matrix Metalloproteinase-9 expression
Tear break-up time | One month
  Non-invasive tear break-up time

CONTACTS AND LOCATIONS:
Overall Officials: Srihari Narayanan, OD, PhD, Principal Investigator — University of the Incarnate Word
Locations (1):
- Rosenberg School of Optometry, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other outside researchers.

REFERENCES:
- [Background] Korb DR, Blackie CA. Debridement-scaling: a new procedure that increases Meibomian gland function and reduces dry eye symptoms. Cornea. 2013 Dec;32(12):1554-7. doi: 10.1097/ICO.0b013e3182a73843. PMID 24145633